CLINICAL TRIAL: NCT02550197
Title: Immunogenicity and Safety of a Quadrivalent Influenza Vaccine Administered Via the Intramuscular Route in Subjects Aged 18 to 60 Years in the Republic of Korea
Brief Title: Immunogenicity and Safety of a Quadrivalent Influenza Vaccine Given by Intramuscular Route in Subjects Aged 18 to 60 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GQM07; U1111-1143-9015 (Other: WHO)
Record Dates: First submitted 2015-09-11; First posted 2015-09-15 (Estimated); Results first posted 2016-11-04 (Estimated); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Influenza
Keywords: Influenza; Quadrivalent influenza vaccine; Trivalent influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- QIV Group (Experimental): Subjects will receive one dose of the Quadrivalent influenza vaccine (QIV) (split virion, inactivated) Northern Hemisphere (NH) 2015-2016 formulation
  Interventions: Biological: Quadrivalent influenza vaccine (QIV) (split virion, inactivated) Northern Hemisphere (NH) 2015-2016
- TIV Group (Active Comparator): Subjects will receive one dose of the Trivalent influenza vaccine (TIV) (split virion, inactivated) NH 2015-2016 formulation
  Interventions: Biological: Trivalent influenza vaccine (TIV) (split virion, inactivated) NH 2015-2016 formulation

INTERVENTIONS:
Biological: Quadrivalent influenza vaccine (QIV) (split virion, inactivated) Northern Hemisphere (NH) 2015-2016 — 0.5 mL, Intramuscular
  Arms: QIV Group
Biological: Trivalent influenza vaccine (TIV) (split virion, inactivated) NH 2015-2016 formulation — 0.5 mL, Intramuscular
  Arms: TIV Group

SUMMARY:
The aim of the trial is to evaluate immunogenicity and safety of the quadrivalent influenza vaccine (QIV) and the trivalent influenza vaccine (TIV) (split-virion inactivated) Northern Hemisphere (NH) 2015 2016 seasonal formulations, in subjects aged 18 to 60 years in the Republic of Korea for the registration of the QIV by the Ministry of Food and Drug Safety.

Objectives:

* To evaluate the immunogenicity of QIV and TIV (split-virion, inactivated) NH 2015-2016 seasonal formulations. The compliance, in terms of immunogenicity, of the QIV NH 2015-2016 formulation, with the requirements of the Committee for Medicinal Products for Human Use (CHMP) Note for Guidance (NfG) CPMP/BWP/214/96 will be assessed.
* To evaluate the safety profile of QIV and TIV (split-virion, inactivated) NH 2015-2016 seasonal formulations

DETAILED DESCRIPTION:
All subjects will receive one dose of either QIV or TIV on Day 0. They will be monitored for safety and immunogenicity for up to Day 21 post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 60 years on the day of inclusion
* Subjects aged 18 years: Assent form has been signed and dated by the subject or by an independent witness, and informed consent form has been signed and dated by at least one parent or another legally acceptable representative or by an independent witness Subjects aged 19 to 60 years: Informed consent form has been signed and dated by the subject or by an independent witness
* Subject and parent/legally acceptable representative (if applicable) are able to attend all scheduled visits and to comply with all trial procedures

Exclusion Criteria:

* Subject is pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination and until at least 3 weeks after vaccination)
* Participation at the time of study enrollment (or in the 4 weeks preceding the trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination or planned receipt of any vaccine until the second visit, 3 weeks following the trial vaccination
* Vaccination against influenza if administered in the context of a clinical trial or a flu vaccination campaign or self-reported history of influenza infection (influenza-like illness) in the previous 6 months
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known history of seropositivity for Human Immunodeficiency Virus (HIV) or Hepatitis C
* Known systemic hypersensitivity to eggs, chicken proteins, neomycin, formaldehyde and octoxynol-9, or to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the study or to a vaccine containing any of the same substances
* Known or suspected thrombocytopenia, contraindicating intramuscular vaccination, based on Investigator's judgment
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination, based on Investigator's judgment
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0°C). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (3):
- South Korea (3):
  - Ansan-si
  - Incheon
  - Seoul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Choi WS, Noh JY, Lee J, Choi JY, Lee JS, Kim MS, Kim HS, Bang J, Lavis N, Kim WJ. Immunogenicity and safety of a split-virion quadrivalent influenza vaccine in adults 18-60 years of age in the Republic of Korea. Hum Vaccin Immunother. 2018 Mar 4;14(3):587-592. doi: 10.1080/21645515.2017.1381808. Epub 2017 Nov 17. PMID 28933625
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 11 September 2015 to 03 November 2015 at 5 clinic sites in the Republic of Korea.
Pre-assignment Details: A total of 300 participants who met all inclusion and no exclusion criteria were enrolled and vaccinated.
Groups:
- Quadrivalent Influenza Vaccine Group: Participants received one dose of the quadrivalent influenza vaccine (QIV) (split virion, inactivated) Northern Hemisphere (NH) 2015-2016 formulation by the intramuscular route.
- Trivalent Influenza Vaccine Group: Participants received one dose of the trivalent influenza vaccine (TIV) (split virion, inactivated) NH 2015-2016 formulation by the Intramuscular route.
Period: Overall Study
Arm/Group | Quadrivalent Influenza Vaccine Group | Trivalent Influenza Vaccine Group
Started | 200 | 100
Completed | 200 | 100
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quadrivalent Influenza Vaccine Group | Trivalent Influenza Vaccine Group | Total
Number analyzed (Participants) | 200 | 100 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 200 | 100 | 300
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age Continuous | 35.9 (9.1) | 35.6 (9.5) | 35.8 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 71 | 221
  Male | 50 | 29 | 79
Region of Enrollment [Number; unit: Participants]
  Korea, Republic of | 200 | 100 | 300

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers of Influenza Antibodies Before and After Vaccination With a Quadrivalent Influenza Vaccine Administered Via the Intramuscular Route
Description: Immunogenicity was evaluated using the hemagglutination inhibition (HAI) technique.
Time Frame: Day 0 (pre-vaccination) and Day 21 post-vaccination
Population: Geometric mean titers of influenza antibodies were assessed in the Immunogenicity Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Arm/Group | Quadrivalent Influenza Vaccine Group | Trivalent Influenza Vaccine Group
Number analyzed (Participants) | 199 | 100
Titers (1/dilution)
  A/H1N1; Day 0 (N=199, 99) | 142 [116 to 174] | 116 [86.1 to 155]
  A/H1N1; Day 21 (N=199, 99) | 583 [516 to 658] | 651 [550 to 771]
  A/H3N2; Day 0 (N=199, 99) | 41.6 [34.1 to 50.9] | 35.8 [27.2 to 47.0]
  A/H3N2; Day 21 (N=199, 99) | 483 [406 to 574] | 691 [543 to 881]
  B/Phuket; Day 0 (N=199, 99) | 256 [212 to 309] | 219 [166 to 290]
  B/Phuket; Day 21 (N=199, 99) | 1068 [950 to 1200] | 1105 [933 to 1308]
  B/Bris; Day 0 (N=199, 100) | 186 [156 to 220] | 139 [107 to 180]
  B/Bris; Day 21 (N=199, 100) | 737 [651 to 835] | 290 [231 to 364]

2. Primary Outcome: Percentage of Participants Achieving Seroprotection Against Influenza Antigens Before and After Vaccination With a Quadrivalent Influenza Vaccine Administered Via the Intramuscular Route
Description: Immunogenicity was evaluated using the hemagglutination inhibition (HAI) technique. Seroprotection was defined as titers ≥ 40 (1/dil) on Day 0 and Day 21.
Time Frame: Day 0 (pre-vaccination) and Day 21 post-vaccination
Population: Seroprotection was assessed in the Immunogenicity Analysis Set.
Measure: Number; unit: Percentage of Participants
Arm/Group | Quadrivalent Influenza Vaccine Group | Trivalent Influenza Vaccine Group
Number analyzed (Participants) | 199 | 100
Percentage of Participants
  A/H1N1; Day 0 (N=199, 99) | 83.4 | 78.8
  A/H1N1; Day 21 (N=199, 99) | 99.5 | 100.0
  A/H3N2; Day 0 (N=199, 99) | 56.3 | 55.6
  A/H3N2; Day 21 (N=199, 99) | 98.0 | 99.0
  B/Phuket; Day 0 (N=199, 99) | 91.5 | 87.9
  B/Phuket; Day 21 (N=199, 99) | 100.0 | 100.0
  B/Bris; Day 0 (N=199, 100) | 89.4 | 85.0
  B/Bris; Day 21 (N=199, 100) | 100.0 | 97.0

3. Primary Outcome: Percentage of Participants With Influenza Antibodies Titers < 10 (1/Dil) Before and After Vaccination With a Quadrivalent Influenza Vaccine Administered Via the Intramuscular Route
Description: Immunogenicity was evaluated using the hemagglutination inhibition (HAI) technique.
Time Frame: Day 0 (pre-vaccination) and Day 21 post-vaccination
Population: Immunogenicity was assessed in the Immunogenicity Analysis Set.
Measure: Number; unit: Percentage of Participants
Arm/Group | Quadrivalent Influenza Vaccine Group | Trivalent Influenza Vaccine Group
Number analyzed (Participants) | 199 | 100
Percentage of Participants
  A/H1N1; Day 0 (N=199, 99) | 5.5 | 6.1
  A/H1N1; Day 21 (N=199, 99) | 0.0 | 0.0
  A/H3N2; Day 0 (N=199, 99) | 17.1 | 20.2
  A/H3N2; Day 21 (N=199, 99) | 0.0 | 0.0
  B/Phuket; Day 0 (N=199, 99) | 1.5 | 1.0
  B/Phuket; Day 21 (N=199, 99) | 0.0 | 0.0
  B/Bris; Day 0 (N=199, 100) | 0.5 | 2.0
  B/Bris; Day 21 (N=199, 100) | 0.0 | 0.0

4. Primary Outcome: Percentage of Participants Achieving Seroconversion or Significant Increase Against Influenza Antigens After Vaccination With a Quadrivalent Influenza Vaccine Administered Via the Intramuscular Route
Description: Immunogenicity was evaluated using the hemagglutination inhibition (HAI) technique. Seroconversion was defined as titers < 10 (1/dil) on Day 0 and post-injection titer ≥ 40 (1/dil) on Day 21, and Significant increase was defined as titers ≥ 10 (1/dil) on Day 0 and ≥ 4-fold increase of post-injection titer on Day 21.
Time Frame: Day 21 post-vaccination
Population: Immunogenicity was assessed in the Immunogenicity Analysis Set.
Measure: Number; unit: Percentage of Participants
Arm/Group | Quadrivalent Influenza Vaccine Group | Trivalent Influenza Vaccine Group
Number analyzed (Participants) | 199 | 100
Percentage of Participants
  A/H1N1 (N=199, 99) | 39.7 | 46.5
  A/H3N2 (N=199, 99) | 72.4 | 84.8
  B/Phuket (N=199, 99) | 48.7 | 53.5
  B/Bris (N=199, 100) | 46.2 | 23.0

5. Primary Outcome: Geometric Mean Titer Ratios of Influenza Virus Antibodies After Vaccination With a Quadrivalent Influenza Vaccine Administered Via the Intramuscular Route
Description: Immunogenicity was evaluated using the hemagglutination inhibition (HAI) technique.
Time Frame: Day 0 (pre-vaccination) and Day 21 post-vaccination
Population: Geometric mean titer ratios of influenza antibodies were assessed in the Immunogenicity Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer ratio
Arm/Group | Quadrivalent Influenza Vaccine Group | Trivalent Influenza Vaccine Group
Number analyzed (Participants) | 199 | 100
Titer ratio
  A/H1N1 (N=199, 99) | 4.10 [3.30 to 5.09] | 5.64 [4.09 to 7.76]
  A/H3N2 (N=199, 99) | 11.6 [9.16 to 14.7] | 19.3 [13.9 to 26.8]
  B/Phuket (N=199, 99) | 4.17 [3.49 to 4.98] | 5.04 [3.81 to 6.67]
  B/Bris (N=199, 100) | 3.97 [3.30 to 4.78] | 2.08 [1.75 to 2.48]

6. Primary Outcome: Percentage of Participants Reporting Solicited Reactions Listed in The Former Committee for Medicinal Products for Human Use Note for Guidance Within 3 Days After Vaccination With a Quadrivalent Influenza Vaccine Administered Via the Intramuscular Route
Description: The solicited reactions evaluated were Injection-site Induration (≥50 mm for at least 4 consecutive days), Injection-site Ecchymosis (injection site bruising), Pyrexia (recorded temperature >38.0˚C for at least 1 day), Malaise, and Shivering (rigors).
Time Frame: Day 0 up Day 3 post-vaccination
Population: Solicited reactions were analyzed in the Safety Analysis Set.
Measure: Number; unit: Percentage of Participants
Arm/Group | Quadrivalent Influenza Vaccine Group | Trivalent Influenza Vaccine Group
Number analyzed (Participants) | 200 | 100
Percentage of Participants
  Reaction listed in the EMA note for guidance | 34.5 | 40.0
  Injection site Induration (≥50 mm for 4 days) | 0.0 | 0.0
  Injection site Ecchymosis (Inj. site Bruising) | 6.0 | 4.0
  Pyrexia (temperature >38.0˚C for at least 1 day) | 0.0 | 0.0
  Malaise | 31.0 | 40.0
  Shivering (Rigors) | 5.5 | 6.0

7. Primary Outcome: Percentage of Participants Reporting Solicited Injection-Site or Systemic Reaction After Vaccination With a Quadrivalent Influenza Vaccine Administered Via the Intramuscular Route
Description: Solicited Injection-site reactions: Pain, Erythema, Swelling, Induration, and Ecchymosis. Solicited Systemic reactions: Fever, Headache, Malaise, Myalgia, and Shivering. Grade 3: Pain, Significant; prevents daily activity; Erythema, Swelling, Induration, and Ecchymosis, >100 mm. Grade 3 Solicited Systemic reactions: Fever, ≥ 39.0˚C; Headache, Malaise, Myalgia, and Shivering, Significant; prevents daily activity.
Time Frame: Day 0 up Day 7 post-vaccination
Population: Solicited injection-site and systemic reactions were analyzed in the Safety Analysis Set.
Measure: Number; unit: Percentage of Participants
Arm/Group | Quadrivalent Influenza Vaccine Group | Trivalent Influenza Vaccine Group
Number analyzed (Participants) | 200 | 100
Percentage of Participants
  Any Injection-site Pain | 70.5 | 64.0
  Grade 3 Injection-site Pain | 1.0 | 0.0
  Any Injection-site Erythema | 2.5 | 3.0
  Grade 3 Injection-site Erythema | 0.0 | 0.0
  Any Injection-site Swelling | 3.5 | 0.0
  Grade 3 Injection-site Swelling | 0.0 | 0.0
  Any Injection-site Induration | 3.0 | 2.0
  Grade 3 Injection-site Induration | 0.0 | 0.0
  Any Injection-site Ecchymosis | 0.0 | 0.0
  Grade 3 Injection-site Ecchymosis | 0.0 | 0.0
  Any Fever | 0.5 | 0.0
  Grade 3 Fever | 0.0 | 0.0
  Any Headache | 16.5 | 20.0
  Grade 3 Headache | 1.5 | 2.0
  Any Malaise | 33.5 | 42.0
  Grade 3 Malaise | 1.5 | 1.0
  Any Myalgia | 51.0 | 49.0
  Grade 3 Myalgia | 1.5 | 0.0
  Any Shivering | 6.5 | 6.0
  Grade 3 Shivering | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 up to Day 21 post-vaccination.
Arm/Group | Quadrivalent Influenza Vaccine Group | Trivalent Influenza Vaccine Group
Serious Adverse Events (participants affected / at risk) | 0/200 | 0/100
Other Adverse Events (participants affected / at risk) | 141/200 | 64/100
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quadrivalent Influenza Vaccine Group (N=200) | Trivalent Influenza Vaccine Group (N=100)
Injection site Pain (General disorders) | 141 (141) | 64 (64)
Headache (Nervous system disorders) | 33 (33) | 20 (20)
Malaise (General disorders) | 67 (67) | 42 (42)
Myalgia (Musculoskeletal and connective tissue disorders) | 102 (102) | 49 (49)
Shivering (General disorders) | 13 (13) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications